CLINICAL TRIAL: NCT02720094
Title: A Phase 2b/3 Double Blind Safety and Efficacy Study of Injectable Cabotegravir Compared to Daily Oral Tenofovir Disoproxil Fumarate/Emtricitabine For Pre-Exposure Prophylaxis in HIV-Uninfected Men and Transgender Women Who Have Sex With Men
Brief Title: Injectable Cabotegravir Compared to TDF/FTC For PrEP in HIV-Uninfected Men and Transgender Women Who Have Sex With Men
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ViiV Healthcare (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPTN 083; 20725 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Results first posted 2023-11-24 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
Keywords: Pre-Exposure Prophylaxis; PrEP
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): In Step 1, participants will receive daily oral CAB and daily oral TDF/FTC placebo for 5 weeks. In Step 2, participants will receive CAB LA and daily oral TDF/FTC placebo to Week 153. In Step 3, participants will receive daily oral TDF/FTC starting at Week 153 and for 48 weeks.
  Interventions: Drug: Cabotegravir Oral Tablet; Drug: TDF/FTC tablets; Drug: Placebo for TDF/FTC tablets; Drug: CAB LA
- Arm B (Experimental): In Step 1, participants will receive daily oral TDF/FTC and daily oral CAB placebo for 5 weeks. In Step 2, participants will receive daily oral TDF/FTC and placebo for CAB LA to Week 153. In Step 3, participants will receive daily oral TDF/FTC starting at Week 153 and for 48 weeks.
  Interventions: Drug: TDF/FTC tablets; Drug: Placebo for cabotegravir oral tablet; Drug: Placebo for CAB LA

INTERVENTIONS:
Drug: Cabotegravir Oral Tablet — 30 mg tablet
  Other Names: Oral cabotegravir
  Arms: Arm A
Drug: TDF/FTC tablets — 300 mg/200 mg fixed-dose combination tablets
  Other Names: Truvada
Drug: Placebo for TDF/FTC tablets
  Other Names: Placebo for Truvada
  Arms: Arm A
Drug: Placebo for cabotegravir oral tablet
  Other Names: Placebo for oral cabotegravir
  Arms: Arm B
Drug: CAB LA — Administered as one 3 mL (600 mg) IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter
  Other Names: Long acting cabotegravir; Injectable cabotegravir
  Arms: Arm A
Drug: Placebo for CAB LA — Administered as one 3 mL IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter
  Other Names: Placebo for long acting cabotegravir
  Arms: Arm B

SUMMARY:
This study will evaluate the safety and efficacy of the injectable drug cabotegravir (CAB LA), for pre-exposure prophylaxis (PrEP) in HIV-uninfected cisgender men and transgender women who have sex with men (MSM and TGW).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of the injectable drug cabotegravir (CAB LA), for pre-exposure prophylaxis (PrEP) in HIV-uninfected cisgender men and transgender women who have sex with men (MSM and TGW).

This study will enroll HIV-uninfected MSM and TGW at risk for acquiring HIV infection. Participants will be followed for a total of 4 years.

This study will take place in three steps. Participants will be randomly assigned to one of two arms:

Arm A:

Step 1: Participants will receive daily oral CAB tablets and daily oral TDF/FTC placebo tablets for 5 weeks.

Step 2: Participants will receive an intramuscular (IM) injection of CAB LA at two time points 4 weeks apart and every 8 weeks thereafter and daily oral TDF/FTC placebo tablets to Week 153.

Arm B:

Step 1: Participants will receive daily oral TDF/FTC tablets and daily oral CAB placebo tablets for 5 weeks.

Step 2: Participants will receive daily oral TDF/FTC tablets and an IM injection of placebo at two time points 4 weeks apart and every 8 weeks thereafter to Week 153.

In Step 3, all participants (Arms A and B) will receive daily oral TDF/FTC tablets starting at Week 153 (last day of Step 2)/Day 0 (first day of Step 3) and continue for 48 weeks.

Participants will attend up to 47 study visits throughout the study. Visits may include physical examinations, blood collection, urine collection, an electrocardiogram (ECG), and rectal swab collection. Some participants may have a bone mineral density-energy x-ray absorptimetry (DXA) scan at select visits.

All participants will be transitioned to locally available HIV prevention services, including services for PrEP, if available, at the end of their participation in the study.

HPTN 083-01 is a sub-study of HPTN 083. The purpose of this study is to evaluate the safety, tolerability, and acceptability of CAB LA for the prevention of HIV among adolescent males. Participants will receive oral CAB for 5 weeks, followed by 29 weeks on CAB LA, then quarterly visits for 48 weeks after final injection. All participants who have received at least one injection will be followed for 48 weeks after their last injection. Total study duration per participant will be approximately 21 months.

HPTN 083-02 is a qualitative sub-study of participants enrolled in HPTN 083. The purpose of this study is to explore potential barriers, facilitators, and potentially modifiable issues related to adherence to clinic visits in the context of injectable PrEP; to learn about preferences and decision making regarding the use of oral versus injectable PrEP, or other biomedical prevention products; and to gather explanatory qualitative data regarding participants' experiences in HPTN 083 to better interpret study results and guide next prevention strategies. Participants in this sub-study will complete one individual semi-structured qualitative interview.

ELIGIBILITY:
Inclusion Criteria:

* MSM and TGW, 18 years or older at the time of screening (male at birth)
* Willing to provide informed consent for the study
* At high risk for sexually acquiring HIV infection based on self-report of at least one of the following:

  * Any condomless receptive anal intercourse in the 6 months prior to enrollment (condomless anal intercourse within a monogamous HIV seronegative concordant relationship does not meet this criterion)
  * More than five partners in the 6 months prior to enrollment (regardless of condom use and HIV serostatus, as reported by the enrollee)
  * Any stimulant drug use in the 6 months prior to enrollment
  * Rectal or urethral gonorrhea or chlamydia or incident syphilis in the 6 months prior to enrollment
  * SexPro score of less than or equal to 16 (U.S. sites only)
* In general good health, as evidenced by the following laboratory values, which must be from specimens obtained within 45 days prior to study enrollment:

  * Non-reactive / negative HIV test results. More information on this criterion can be found in the protocol.
  * Hemoglobin greater than 11 g/dL,
  * Absolute neutrophil count greater than 750 cells/mm^3
  * Platelet count greater than or equal to 100,000/mm^3
  * Calculated creatinine clearance greater than or equal to 60 mL/minute using the Cockcroft-Gault equation (use sex at birth for calculation)

    * Although not protocol exclusionary, sites should carefully consider the advisability of enrolling participants with calculated creatinine clearance between 60-70 mL/min, as limited changes in creatinine clearance during study conduct will lead to protocol-mandated product holds and may alter the risk-benefit considerations of study participation
  * Alanine aminotransferase (ALT) less than 2 times the upper limit of normal (ULN)
  * Total bilirubin less than or equal to 2.5 times ULN
  * Hepatitis B virus (HBV) surface antigen (HBsAg) negative
  * Hepatitis C virus (HCV) Ab negative
  * No Grade 3 or higher laboratory abnormalities on any laboratory tests obtained at screening, including tests obtained as part of a panel of tests ordered to obtain the protocol-required laboratory test results.
* No medical condition that, in the opinion of the study investigator, would interfere with the conduct of the study (e.g., provided by self-report, or found upon medical history and examination or in available medical records)
* Willing to undergo all required study procedures

Exclusion Criteria:

* One or more reactive or positive HIV test result at Screening or Enrollment, even if HIV infection is not confirmed
* Active or recent use of any illicit intravenous drugs ("recent" defined as in the 90 days prior to enrollment)
* Co-enrollment in any other interventional research study or other concurrent studies that may interfere with this study (as provided by self-report or other available documentation. Exceptions may be made if appropriate after consultation with the CMC.)
* Past or current participation in HIV vaccine trial. An exception will be made for participants that can provide documentation of receipt of placebo (not active arm). Note: Past participation in a monoclonal antibody study is not exclusionary, effective as of Version 1.0 of HPTN 083.
* Clinically significant cardiovascular disease, as defined by history/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease
* Inflammatory skin conditions that compromise the safety of intramuscular (IM) injections, per the discretion of the Investigator of Record. Mild skin conditions may not be exclusionary at the discretion of the Investigator of Record (IoR) or designee in consultation with the CMC
* Has a tattoo or other dermatological condition overlying the buttock region which in the opinion of the IoR or designee, in consultation with the CMC, may interfere with interpretation of injection site reactions
* Current or chronic history of liver disease (e.g., non-alcoholic or alcoholic steatohepatitis) or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome, asymptomatic gallstones, or cholecystectomy)
* Coagulopathy (primary or iatrogenic) which would contraindicate IM injection (concomitant anticoagulant or anti-platelet therapy use should be discussed with the CMC)
* Active or planned use of prohibited medications as described in the Investigator's Brochure or listed in the Study Specific Procedures (SSP) Manual (provided by self-report, or obtained from medical history or medical records). In particular, future use of TDF/FTC at any point during the study.
* Known or suspected allergy to study product components (active or placebo), including egg or soy products (egg and soy products are contained in Intralipid)
* Surgically-placed or injected buttock implants or fillers, per self-report. Contact the CMC for guidance regarding questions about individual cases.
* Alcohol or substance use that, in the opinion of the study investigator, would jeopardize the safety of the participant on study (e.g., provided by self-report, or found upon medical history and examination or in available medical records).
* History of seizure disorder, per self-report
* QTc interval (B or F) greater than 500 msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4570 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael J. Landovitz, MD, MSc, Study Chair — University of California, Los Angeles
Locations (43):
- United States (27):
  - Alabama CRS, Birmingham, Alabama
  - UCLA Vine Street Clinic CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - East Bay AIDS Center (EBAC) CRS, Oakland, California
  - Bridge HIV CRS, San Francisco, California
  - Children's Hospital Colorado CRS, Aurora, Colorado
  - George Washington Univ. CRS, Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Adolescent & Young Adult Research at The CORE Center (AYAR at CORE), Chicago, Illinois
  - UIC Project WISH CRS, Chicago, Illinois
  - New Orleans Adolescent Trials Unit CRS, New Orleans, Louisiana
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Harlem Prevention Center CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - Bronx Prevention Research Center CRS, The Bronx, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Houston AIDS Research Team CRS, Houston, Texas
- Argentina (2):
  - Hospital General de Agudos JM Ramos Mejía CRS, Ciudad de Buenos Aires, Buenos Aires
  - Fundacion Huesped CRS, Buenos Aires
- Brazil (4):
  - Hospital Nossa Senhora da Conceicao CRS, Porto Alegre, Rio Grande do Sul
  - Centro de Referencia e Treinamento DST/AIDS CRS, São Paulo, São Paulo
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
  - Centro de Pesquisas Clínicas IC-HCFMUSP CRS, São Paulo
- Peru (5):
  - ACSA CRS, Iquitos, Maynas
  - CITBM - UNIDEC, Centro de Investigaciones Tecnológicas, Biomédicas y Medioambientales CRS, Bellavista, Provincia Constitucional del Callao
  - Via Libre CRS, Lima
  - Barranco CRS, Lima
  - San Miguel CRS, Lima
- Groote Schuur HIV CRS, Cape Town, Western Cape, South Africa
- Thailand (3):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Pathum Wan, Bangkok
  - Silom Community Clinic CRS, Bangkok, Changwat Nonthaburi
  - CMU HIV Prevention CRS, Chiang Mai
- Yen Hoa Health Clinic CRS, Hanoi, Vietnam

REFERENCES:
- [Derived] Brown TT, Arao RF, Warsi M, Phanuphak N, Vasconcelos R, Oyedele T, Sullivan PA, Hanscom B, Rooney JF, Rinehart AR, McCauley M, Grinsztejn B, Landovitz RJ. Bone Changes With Long-Acting Cabotegravir or Tenofovir Disoproxil Fumarate/Emtricitabine for HIV Prevention in Cisgender Men and Transgender Women: HPTN 083. Clin Infect Dis. 2025 Dec 24;81(5):983-986. doi: 10.1093/cid/ciaf221. PMID 40590452
- [Derived] Psaros C, Goodman GR, Lee JS, Rice W, Kelley CF, Oyedele T, Coelho LE, Phanuphak N, Singh Y, Middelkoop K, Griffith S, McCauley M, Rooney J, Rinehart AR, Clark J, Go V, Sugarman J, Fields SD, Adeyeye A, Grinsztejn B, Landovitz RJ, Safren SA; HPTN 083-02 Study Team. HPTN 083-02: factors influencing adherence to injectable PrEP and retention in an injectable PrEP study. J Int AIDS Soc. 2024 May;27(5):e26252. doi: 10.1002/jia2.26252. PMID 38783534
- [Derived] Han K, Patel P, McCallister S, Rinehart AR, Gandhi Y, Spreen W, Landovitz RJ, Delany-Moretlwe S, Marzinke MA, McKeon T, Budnik P, van Wyk J, Ford SL. Long-acting cabotegravir pharmacokinetics with and without oral lead-in for HIV PrEP. Antimicrob Agents Chemother. 2024 Jun 5;68(6):e0147523. doi: 10.1128/aac.01475-23. Epub 2024 May 6. PMID 38709006
- [Derived] Landovitz RJ, Hanscom BS, Clement ME, Tran HV, Kallas EG, Magnus M, Sued O, Sanchez J, Scott H, Eron JJ, Del Rio C, Fields SD, Marzinke MA, Eshleman SH, Donnell D, Spinelli MA, Kofron RM, Berman R, Piwowar-Manning EM, Richardson PA, Sullivan PA, Lucas JP, Anderson PL, Hendrix CW, Adeyeye A, Rooney JF, Rinehart AR, Cohen MS, McCauley M, Grinsztejn B; HPTN 083 Study Team. Efficacy and safety of long-acting cabotegravir compared with daily oral tenofovir disoproxil fumarate plus emtricitabine to prevent HIV infection in cisgender men and transgender women who have sex with men 1 year after study unblinding: a secondary analysis of the phase 2b and 3 HPTN 083 randomised controlled trial. Lancet HIV. 2023 Dec;10(12):e767-e778. doi: 10.1016/S2352-3018(23)00261-8. Epub 2023 Nov 9. PMID 37952550
- [Derived] Marzinke MA, Hanscom B, Wang Z, Safren SA, Psaros C, Donnell D, Richardson PA, Sullivan P, Eshleman SH, Jennings A, Feliciano KG, Jalil E, Coutinho C, Cardozo N, Maia B, Khan T, Singh Y, Middelkoop K, Franks J, Valencia J, Sanchez N, Lucas J, Rooney JF, Rinehart AR, Ford S, Adeyeye A, Cohen MS, McCauley M, Landovitz RJ, Grinsztejn B; HPTN 083 study group. Efficacy, safety, tolerability, and pharmacokinetics of long-acting injectable cabotegravir for HIV pre-exposure prophylaxis in transgender women: a secondary analysis of the HPTN 083 trial. Lancet HIV. 2023 Nov;10(11):e703-e712. doi: 10.1016/S2352-3018(23)00200-X. Epub 2023 Sep 29. PMID 37783219
- [Derived] Landovitz RJ, Donnell D, Clement ME, Hanscom B, Cottle L, Coelho L, Cabello R, Chariyalertsak S, Dunne EF, Frank I, Gallardo-Cartagena JA, Gaur AH, Gonzales P, Tran HV, Hinojosa JC, Kallas EG, Kelley CF, Losso MH, Madruga JV, Middelkoop K, Phanuphak N, Santos B, Sued O, Valencia Huamani J, Overton ET, Swaminathan S, Del Rio C, Gulick RM, Richardson P, Sullivan P, Piwowar-Manning E, Marzinke M, Hendrix C, Li M, Wang Z, Marrazzo J, Daar E, Asmelash A, Brown TT, Anderson P, Eshleman SH, Bryan M, Blanchette C, Lucas J, Psaros C, Safren S, Sugarman J, Scott H, Eron JJ, Fields SD, Sista ND, Gomez-Feliciano K, Jennings A, Kofron RM, Holtz TH, Shin K, Rooney JF, Smith KY, Spreen W, Margolis D, Rinehart A, Adeyeye A, Cohen MS, McCauley M, Grinsztejn B; HPTN 083 Study Team. Cabotegravir for HIV Prevention in Cisgender Men and Transgender Women. N Engl J Med. 2021 Aug 12;385(7):595-608. doi: 10.1056/NEJMoa2101016. PMID 34379922
- [Derived] Scarsi KK. Chasing the cabotegravir tail: implications for prevention. Lancet HIV. 2020 Jul;7(7):e451-e453. doi: 10.1016/S2352-3018(20)30165-X. Epub 2020 Jun 1. No abstract available. PMID 32497490

RESULTS

PARTICIPANT FLOW:
Groups:
- Cabotegravir: In Step 1, participants will receive daily oral cabotegravir (CAB) and daily oral Tenofovir/emtricitabine (TDF/FTC) placebo for 5 weeks. In Step 2, participants will receive long-acting injectable cabotegravir (CAB LA) and daily oral TDF/FTC placebo to Week 153. In Step 3, participants will receive daily oral TDF/FTC starting at Week 153 and for 48 weeks.
  Cabotegravir tablets: 30 mg tablets
  TDF/FTC tablets: 300 mg/200 mg fixed-dose combination tablets
  TDF/FTC placebo tablets
  CAB LA: Administered as one 3 mL (600 mg) IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter
- TDF/FTC: In Step 1, participants will receive daily oral Tenofovir/emtricitabine (TDF/FTC) and daily oral cabotegravir (CAB) placebo for 5 weeks. In Step 2, participants will receive daily oral TDF/FTC and placebo for long-acting injectable cabotegravir (CAB LA) to Week 153. In Step 3, participants will receive daily oral TDF/FTC starting at Week 153 and for 48 weeks.
  TDF/FTC tablets: 300 mg/200 mg fixed-dose combination tablets
  CAB placebo tablets
  Placebo for CAB LA: Administered as one 3 mL IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter
Period: Overall Study
Arm/Group | Cabotegravir | TDF/FTC
Started | 2283 | 2287
Ongoing (Ongoing in the study indicates the participant has not terminated study.) | 2210 | 2203
Terminated From the Study (Excludes participants who completed the study.) | 67 | 78
Completed (Completed the study indicates a participant has seroconverted or has entered Step 3 after reaching Week 145 visit and was subsequently followed for 48 weeks in Step 3 without prior IP discontinuation or study termination or has entered Step 3 after discontinuation of IP and was subsequently followed for 48 weeks and was followed for a total of 3 years from enrollment.) | 7 | 6
Not Completed | 2276 | 2281
Not completed — Ongoing | 2210 | 2203
Not completed — Scheduled exit visit/end of study | 2 | 1
Not completed — Death | 4 | 7
Not completed — Withdrawal by Subject | 55 | 56
Not completed — Lost to Follow-up | 2 | 7
Not completed — Physician Decision | 1 | 3
Not completed — Inappropriate enrollment | 1 | 3
Not completed — Relocation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cabotegravir: In Step 1, participants will receive daily oral CAB and daily oral TDF/FTC placebo for 5 weeks. In Step 2, participants will receive CAB LA and daily oral TDF/FTC placebo to Week 153. In Step 3, participants will receive daily oral TDF/FTC starting at Week 153 and for 48 weeks.
  Cabotegravir tablets: 30 mg tablets
  TDF/FTC tablets: 300 mg/200 mg fixed-dose combination tablets
  TDF/FTC placebo tablets
  CAB LA: Administered as one 3 mL (600 mg) IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter
- TDF/FTC: In Step 1, participants will receive daily oral TDF/FTC and daily oral CAB placebo for 5 weeks. In Step 2, participants will receive daily oral TDF/FTC and placebo for CAB LA to Week 153. In Step 3, participants will receive daily oral TDF/FTC starting at Week 153 and for 48 weeks.
  TDF/FTC tablets: 300 mg/200 mg fixed-dose combination tablets
  CAB placebo tablets
  Placebo for CAB LA: Administered as one 3 mL IM injection in the gluteal muscle at two time points 4 weeks apart and every 8 weeks thereafter
- Total: Total of all reporting groups
Arm/Group | Cabotegravir | TDF/FTC | Total
Number analyzed (Participants) | 2283 | 2287 | 4570
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (8.17) | 28.2 (8.14) | 28.1 (8.15)
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [22 to 32] | 26 [22 to 32] | 26 [22 to 32]
Age, Customized [Count of Participants; unit: Participants]
  18-24 years | 931 | 915 | 1846
  25-34 years | 940 | 931 | 1871
  35-44 years | 285 | 313 | 598
  45-54 years | 103 | 109 | 212
  55-60 years | 19 | 17 | 36
  61+ years | 5 | 2 | 7
Age, Customized [Count of Participants; unit: Participants]
  <30 years | 1572 | 1510 | 3082
  >=30 years | 711 | 777 | 1488
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Men who have sex with men | 2014 | 1982 | 3996
  Transgender women | 266 | 304 | 570
  Prefer not to answer | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity categories as defined by the National Institutes of Health and the Office of Management and Budget
  Participants
    Hispanic or Latino | 1043 | 1067 | 2110
    Not Hispanic or Latino | 1240 | 1219 | 2459
    Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 616 | 600 | 1216
  Asian | 417 | 406 | 823
  Native Hawaiian or Other Pacific Islander | 5 | 2 | 7
  Black or African American | 565 | 569 | 1134
  White | 618 | 649 | 1267
  More than one race | 49 | 54 | 103
  Unknown or Not Reported | 13 | 7 | 20
Region of Enrollment [Number; unit: participants] — Geographical regions and their representative countries are classified as: United States (U.S.), Latin America (Argentina, Brazil and Peru), Asia (Vietnam and Thailand), Africa (South Africa)
  participants
    Argentina | 169 | 168 | 337
    Vietnam | 100 | 99 | 199
    United States | 850 | 851 | 1701
    Brazil | 395 | 401 | 796
    Africa | 78 | 74 | 152
    Thailand | 275 | 278 | 553
    Peru | 416 | 416 | 832
Marital Status [Count of Participants; unit: Participants]
  Married/Civil Union/Legal Partnership | 79 | 98 | 177
  Living with Primary or Main Partner | 138 | 154 | 292
  Have Primary or Main Partner, not Living Together | 171 | 165 | 336
  Single/Divorced/Widowed | 1889 | 1865 | 3754
  Other | 6 | 5 | 11
Education [Count of Participants; unit: Participants]
  No Schooling | 2 | 6 | 8
  Primary School, not complete | 12 | 17 | 29
  Primary School, complete | 16 | 25 | 41
  Secondary School, not complete | 119 | 113 | 232
  Secondary School, complete | 371 | 410 | 781
  Technical Training, not complete | 74 | 79 | 153
  Technical Training, complete | 113 | 109 | 222
  College/University or Higher, not complete | 708 | 712 | 1420
  College/University or Higher, complete | 868 | 816 | 1684

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Documented Incident HIV Infections During Steps 1 and 2
Description: All HIV infections included in this analysis have been reviewed and confirmed by an independent, blinded Endpoint Adjudication Committee (EAC).
Time Frame: HIV tests at enrollment, weeks 2, 4, 5, every injection visit (every 8 weeks) and every safety visit (2 weeks after each injection visit). Analyzed through week 153 or the date of DSMB decision to unblind all participants, whichever is earliest.
Population: mITT Population (Steps 1 and 2): Participants who were inappropriately enrolled are excluded. Participants who were found by the EAC to be HIV infected at enrollment are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 2280 | 2281
Participants | 13 | 39
Statistical Analysis 1: Comparison: Cabotegravir vs TDF/FTC; Test type: Superiority; p = 0.0005, Regression, Cox; A bias-adjusted hazard ratio = 0.340, 95% CI 2-sided [0.18 to 0.62] — The bias-adjusted hazard ratio, CI, and p-value account for the group-sequential trial design and the early stopping time
Statistical Analysis 2: Comparison: Cabotegravir vs TDF/FTC; Test type: Superiority; p = 0.0005, Regression, Cox; Hazard Ratio (HR) = 0.328, 95% CI 2-sided [0.18 to 0.61] — The unadjusted hazard ratio is based on a Cox proportional hazards model stratified by region

2. Primary Outcome: Number of Participants Experiencing Grade 2 or Higher Clinical and Laboratory Adverse Events
Description: The primary safety endpoint analyses included Grade 2 or higher clinical and laboratory AEs during Steps 1 and 2.
Time Frame: Treatment emergent AE* measured with onset date through participant's last study visit, or the date of DSMB decision to unblind all participants, whichever is earliest. Assessed at each visit (injections visits q 8 weeks and safety visits q 8 weeks).
Population: Inappropriately enrolled participants, participants with invalid ID due to duplicate screening or enrollment and participants who did not receive any oral study drug are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 2280 | 2282
Participants | 2106 | 2116

3. Secondary Outcome: Number of Participants With Documented Incident HIV Infections in Step 2
Description: Evaluate incident HIV-1infections occurring only during Step 2, using the Injection Step 2 Efficacy population
Time Frame: as for outcome 1
Population: Injection step 2 efficacy: The subgroup of the mITT population who received at least one injection and had at least one HIV result assessed after the first injection visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 2114 | 2079
Participants | 8 | 37
Statistical Analysis 1: Comparison: Cabotegravir vs TDF/FTC; The analysis population Injection Step 2 Efficacy consists of the subset of the mITT population who received at least one injection and had at least one HIV test result after the week 5 injection visit; Test type: Superiority; p < 0.001, Regression, Cox — The P-Values are two-sided; Hazard Ratio (HR) = 0.210, 95% CI 2-sided [0.10 to 0.45]

4. Secondary Outcome: Changes From Baseline in Creatinine and Creatinine Clearance Levels
Description: Change from baseline at each visit is the difference between the creatine (and creatinine clearance) value as measured on the date of visit, compared to the value as measured at the enrollment visit.
Time Frame: Reported week 57 (injection visit #8) and week 105 (injection visit #14)
Population: All subjects who received at least one dose of study product, and for whom have results for creatine and creatinine clearance at enrollment AND for at least one of the following two time points: Week 57 and Week 105.
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 1364 | 1360
umol/L
  Week 57 (Injection #8) | 0.90 [-5.30 to 7.10] | 1.70 [-4.40 to 7.90]
  Week 105 (Injection #14): number analyzed (Participants) | 466 | 484
  Week 105 (Injection #14) | 0.90 [-5.30 to 8.80] | 2.30 [-3.50 to 8.80]

5. Secondary Outcome: Number of Participants With Grade 3 or 4 Liver-related Adverse Events (AEs)
Description: Laboratory assessment of alanine aminotransferase (ALT), aspartate aminotransferase (AST), TBili, creatine phosphokinase (CPK), or clinical assessment of jaundice/icterus.
Time Frame: Treatment emergent AE measured with onset date through participant's last study visit, or the date of DSMB decision to unblind all participants, whichever is first. Assessed at each visit. (Injection visits q 8 weeks and safety visits q 8 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 2280 | 2282
Participants | 73 | 96

6. Secondary Outcome: Incidence of Resistance Mutations to Study Products (Including But Not Limited to K65R, M184V/I, Q148R) Among Seroconverters
Description: Frequency of the detection of specific viral mutations known to confer resistance to specific classes of antiviral drugs as identified in specimens collected from infected participants during follow-up after HIV infection.
Time Frame: Measured from date of detection of infection, up to 4 years after study entry, with timing/intervals as determined by the HPTN laboratory center
Population: All participants in the mITT population who acquired HIV, including those who were found to have acquired HIV prior to randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 14 | 42
Participants
  Any resistance | 8 | 13
  PI resistance | 0 | 0
  NNRTI resistance | 3 | 10
  NRTI resistance | 1 | 6
  INSTI resistance | 6 | 0

7. Secondary Outcome: Changes in Weight From Baseline
Description: Change in weight from baseline is the difference between the weight (kg) as collected at each study visit and the weight collected at the enrollment visit.
Time Frame: Reported through the week 153 injection, or the date of DSMB decision to unblind all participants, whichever is earliest. Collected at each injection visit (every 8 weeks).
Population: Enrolled participants with available data at each visit
Measure: Median (Inter-Quartile Range); unit: Kg
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 2282 | 2284
Kg
  Week 5 (Injection #1): number analyzed (Participants) | 2108 | 2078
  Week 5 (Injection #1) | 0.4 [-0.7 to 1.5] | 0.1 [-1.0 to 1.1]
  Week 9 (Injection #2): number analyzed (Participants) | 2038 | 2012
  Week 9 (Injection #2) | 0.5 [-0.9 to 1.8] | 0.0 [-1.3 to 1.3]
  Week 17 (Injection #3): number analyzed (Participants) | 1941 | 1943
  Week 17 (Injection #3) | 0.7 [-0.9 to 2.4] | 0.0 [-1.7 to 1.6]
  Week 25 (Injection #4): number analyzed (Participants) | 1876 | 1875
  Week 25 (Injection #4) | 0.9 [-1.0 to 2.7] | -0.2 [-2.0 to 1.8]
  Week 33 (Injection #5): number analyzed (Participants) | 1764 | 1765
  Week 33 (Injection #5) | 1.0 [-1.0 to 3.1] | 0.0 [-2.2 to 1.9]
  Week 41 (Injection #6): number analyzed (Participants) | 1625 | 1613
  Week 41 (Injection #6) | 1.2 [-1.0 to 3.5] | 0.0 [-2.1 to 2.4]
  Week 49 (Injection #7): number analyzed (Participants) | 1467 | 1464
  Week 49 (Injection #7) | 1.5 [-0.9 to 3.8] | 0.0 [-2.3 to 2.6]
  Week 57 (Injection #8): number analyzed (Participants) | 1362 | 1361
  Week 57 (Injection #8) | 1.2 [-1.2 to 4.0] | 0.2 [-2.5 to 2.5]
  Week 65 (Injection #9): number analyzed (Participants) | 1207 | 1197
  Week 65 (Injection #9) | 1.7 [-0.9 to 4.5] | 0.5 [-2.4 to 3.1]
  Week #73 (Injection #10): number analyzed (Participants) | 1038 | 1037
  Week #73 (Injection #10) | 1.8 [-0.9 to 5.0] | 0.5 [-2.3 to 3.3]
  Week 81 (Injection #11): number analyzed (Participants) | 881 | 905
  Week 81 (Injection #11) | 2.0 [-1.0 to 5.2] | 0.5 [-2.3 to 3.9]
  Week 89 (Injection #12): number analyzed (Participants) | 747 | 761
  Week 89 (Injection #12) | 2.2 [-0.9 to 5.8] | 0.5 [-2.3 to 3.9]
  Week 97 (Injection #13): number analyzed (Participants) | 603 | 600
  Week 97 (Injection #13) | 2.1 [-0.9 to 5.9] | 1.0 [-1.9 to 4.0]
  Week #105 (Injection #14): number analyzed (Participants) | 464 | 483
  Week #105 (Injection #14) | 2.1 [-1.0 to 6.3] | 0.9 [-2.0 to 4.8]
  Week 113 (Injection #15): number analyzed (Participants) | 376 | 374
  Week 113 (Injection #15) | 2.6 [-0.5 to 7.2] | 1.4 [-2.3 to 5.3]
  Week 121 (Injection #16): number analyzed (Participants) | 298 | 291
  Week 121 (Injection #16) | 2.8 [-0.8 to 7.2] | 1.0 [-2.5 to 5.1]
  Week 129 (Injection #17): number analyzed (Participants) | 234 | 220
  Week 129 (Injection #17) | 2.9 [-0.9 to 7.1] | 1.3 [-2.1 to 4.8]
  Week 137 (Injection #18): number analyzed (Participants) | 169 | 148
  Week 137 (Injection #18) | 2.7 [-1.0 to 7.8] | 1.2 [-2.5 to 5.2]
  Week 145 (Injection #19): number analyzed (Participants) | 112 | 91
  Week 145 (Injection #19) | 2.7 [-1.4 to 7.3] | 1.9 [-1.9 to 5.4]
  Week 153 (Injection #20): number analyzed (Participants) | 59 | 55
  Week 153 (Injection #20) | 2.9 [-0.2 to 7.5] | 0.7 [-2.0 to 6.4]

8. Secondary Outcome: Changes in Systolic Blood Pressure From Baseline
Description: Change in blood pressure from baseline is the difference between the blood pressure as collected at each study visit and the blood pressure collected at the enrollment visit. Reported in separate tables for systole and diastole.
Time Frame: Reported through the week 153 injection, or the date of DSMB decision to unblind all participants, whichever is earliest. Assessed at each injection visit (every 8 weeks).
Population: Includes the subset of subjects who received any study product, including those were subsequently deemed to be inappropriately enrolled.
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 2281 | 2285
mmHg
  Week 5 (Injection #1): number analyzed (Participants) | 2110 | 2074
  Week 5 (Injection #1) | 0.0 [-8.0 to 7.0] | 0.0 [-8.0 to 7.0]
  Week 9 (Injection #2): number analyzed (Participants) | 2038 | 2011
  Week 9 (Injection #2) | 0.0 [-9.0 to 7.0] | -1.0 [-9.0 to 6.0]
  Week 17 (Injection #3): number analyzed (Participants) | 1938 | 1943
  Week 17 (Injection #3) | 0.0 [-8.0 to 7.0] | 0.0 [-9.0 to 7.0]
  Week 25 (Injection #4): number analyzed (Participants) | 1875 | 1874
  Week 25 (Injection #4) | 0.0 [-8.0 to 7.0] | 0.0 [-9.0 to 7.0]
  Week 33 (Injection #5): number analyzed (Participants) | 1761 | 1764
  Week 33 (Injection #5) | 0.0 [-8.0 to 8.0] | 0.0 [-9.0 to 6.0]
  Week 41 (Injection #6): number analyzed (Participants) | 1623 | 1609
  Week 41 (Injection #6) | 0.0 [-9.0 to 8.0] | 0.0 [-8.0 to 7.0]
  Week 49 (Injection #7): number analyzed (Participants) | 1465 | 1464
  Week 49 (Injection #7) | 0.0 [-9.0 to 8.0] | 0.0 [-9.0 to 7.0]
  Week 57 (Injection #8): number analyzed (Participants) | 1360 | 1359
  Week 57 (Injection #8) | 0.0 [-8.0 to 8.0] | -1.0 [-10.0 to 6.0]
  Week 65 (Injection #9): number analyzed (Participants) | 1207 | 1195
  Week 65 (Injection #9) | 0.0 [-8.0 to 7.0] | 0.0 [-9.0 to 7.0]
  Week 73 (Injection #10): number analyzed (Participants) | 1035 | 1036
  Week 73 (Injection #10) | 0.0 [-8.0 to 9.0] | 0.0 [-8.0 to 7.0]
  Week 81 (Injection #11): number analyzed (Participants) | 879 | 902
  Week 81 (Injection #11) | 0.5 [-8.0 to 9.0] | 0.0 [-8.0 to 8.0]
  Week 89 (Injection #12): number analyzed (Participants) | 747 | 759
  Week 89 (Injection #12) | 0.0 [-8.0 to 9.0] | -1.0 [-9.0 to 7.0]
  Week 97 (Injection #13): number analyzed (Participants) | 602 | 600
  Week 97 (Injection #13) | 1.0 [-7.0 to 9.0] | 0.0 [-8.0 to 7.0]
  Week 105 (Injection #14): number analyzed (Participants) | 462 | 482
  Week 105 (Injection #14) | 1.0 [-7.0 to 9.0] | 0.0 [-8.0 to 8.0]
  Week 113 (Injection #15): number analyzed (Participants) | 376 | 374
  Week 113 (Injection #15) | 0.0 [-6.0 to 8.0] | 0.0 [-8.0 to 8.0]
  Week 121 (Injection #16): number analyzed (Participants) | 298 | 290
  Week 121 (Injection #16) | 1.0 [-7.0 to 8.0] | 0.0 [-8.0 to 9.0]
  Week 129 (Injection #17): number analyzed (Participants) | 233 | 219
  Week 129 (Injection #17) | 2.0 [-7.0 to 10.0] | 2.0 [-6.5 to 11.0]
  Week 137 (Injection #18): number analyzed (Participants) | 168 | 148
  Week 137 (Injection #18) | 0.0 [-7.0 to 9.0] | 2.0 [-8.0 to 10.0]
  Week 145 (Injection #19): number analyzed (Participants) | 112 | 91
  Week 145 (Injection #19) | 1.0 [-7.0 to 11.0] | 3.5 [-8.0 to 10.0]
  Week 153 (Injection #20): number analyzed (Participants) | 59 | 55
  Week 153 (Injection #20) | 2.0 [-4.0 to 9.0] | 2.0 [-9.0 to 13.0]

9. Secondary Outcome: Changes in Diastolic Blood Pressure From Baseline
Description: as for outcome 8
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 2281 | 2285
mmHg
  Week 5 (Injection #1): number analyzed (Participants) | 2110 | 2074
  Week 5 (Injection #1) | 0.0 [-7.0 to 5.0] | -1.0 [-7.0 to 4.0]
  Week 9 (Injection #2): number analyzed (Participants) | 2038 | 2011
  Week 9 (Injection #2) | 0.0 [-7.0 to 4.0] | 0.0 [-7.0 to 5.0]
  Week 17 (Injection #3): number analyzed (Participants) | 1938 | 1943
  Week 17 (Injection #3) | 0.0 [-7.0 to 5.0] | 0.0 [-7.0 to 5.0]
  Week 25 (Injection #4): number analyzed (Participants) | 1875 | 1873
  Week 25 (Injection #4) | 0.0 [-7.0 to 5.0] | 0.0 [-7.0 to 5.0]
  Week 33 (Injection #5): number analyzed (Participants) | 1761 | 1764
  Week 33 (Injection #5) | 0.0 [-7.0 to 6.0] | 0.0 [-7.0 to 5.0]
  Week 41 (Injection #6): number analyzed (Participants) | 1623 | 1609
  Week 41 (Injection #6) | 0.0 [-7.0 to 5.0] | -1.0 [-7.0 to 5.0]
  Week 49 (Injection #7): number analyzed (Participants) | 1465 | 1464
  Week 49 (Injection #7) | 0.0 [-7.0 to 5.0] | -1.0 [-7.0 to 5.0]
  Week 57 (Injection #8): number analyzed (Participants) | 1360 | 1359
  Week 57 (Injection #8) | 0.0 [-6.0 to 6.0] | 0.0 [-7.0 to 6.0]
  Week 65 (Injection #9): number analyzed (Participants) | 1207 | 1195
  Week 65 (Injection #9) | 0.0 [-7.0 to 5.0] | 0.0 [-7.0 to 6.0]
  Week 73 (Injection #10): number analyzed (Participants) | 1035 | 1036
  Week 73 (Injection #10) | 0.0 [-6.0 to 5.0] | 0.0 [-7.0 to 6.0]
  Week 81 (Injection #11): number analyzed (Participants) | 879 | 902
  Week 81 (Injection #11) | 0.0 [-6.0 to 6.0] | -1.0 [-7.0 to 5.0]
  Week 89 (Injection #12): number analyzed (Participants) | 747 | 759
  Week 89 (Injection #12) | 0.0 [-7.0 to 5.0] | -1.0 [-6.0 to 5.0]
  Week 97 (Injection #13): number analyzed (Participants) | 602 | 600
  Week 97 (Injection #13) | 0.0 [-7.0 to 6.0] | -1.0 [-8.0 to 5.0]
  Week 105 (Injection #14): number analyzed (Participants) | 462 | 482
  Week 105 (Injection #14) | 0.5 [-6.0 to 7.0] | 0.0 [-6.0 to 6.0]
  Week 113 (Injection #15): number analyzed (Participants) | 376 | 374
  Week 113 (Injection #15) | 1.0 [-6.0 to 7.0] | 0.0 [-6.0 to 7.0]
  Week 121 (Injection #16): number analyzed (Participants) | 298 | 290
  Week 121 (Injection #16) | 0.0 [-6.0 to 6.5] | -1.0 [-7.0 to 6.0]
  Week 129 (Injection #17): number analyzed (Participants) | 233 | 219
  Week 129 (Injection #17) | 1.0 [-6.0 to 9.0] | 0.0 [-7.0 to 5.0]
  Week 137 (Injection #18): number analyzed (Participants) | 168 | 148
  Week 137 (Injection #18) | 0.0 [-5.0 to 7.0] | 0.0 [-6.0 to 5.0]
  Week 145 (Injection #19): number analyzed (Participants) | 112 | 91
  Week 145 (Injection #19) | 1.0 [-5.0 to 8.0] | -2.0 [-6.0 to 5.0]
  Week 153 (Injection #20): number analyzed (Participants) | 59 | 55
  Week 153 (Injection #20) | 2.5 [-6.0 to 8.0] | 0.0 [-4.0 to 4.0]

10. Secondary Outcome: Changes in Pulse Rate From Baseline
Description: Change in pulse rate from baseline is the difference between the pulse rate as collected at each study visit and the pulse rate collected at the enrollment visit.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: beats/min
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 2281 | 2285
beats/min
  Week 5 (Injection #1): number analyzed (Participants) | 2110 | 2075
  Week 5 (Injection #1) | 2.0 [-4.0 to 9.0] | 1.0 [-5.0 to 8.0]
  Week 9 (Injection #2): number analyzed (Participants) | 2038 | 2010
  Week 9 (Injection #2) | 2.0 [-5.0 to 9.0] | 1.0 [-5.0 to 8.0]
  Week 17 (Injection #3): number analyzed (Participants) | 1937 | 1945
  Week 17 (Injection #3) | 2.0 [-5.0 to 9.0] | 2.0 [-5.0 to 9.0]
  Week 25 (Injection #4): number analyzed (Participants) | 1873 | 1873
  Week 25 (Injection #4) | 2.0 [-5.0 to 9.0] | 2.0 [-5.0 to 9.0]
  Week 33 (Injection #5): number analyzed (Participants) | 1761 | 1764
  Week 33 (Injection #5) | 3.0 [-5.0 to 10.0] | 2.0 [-5.0 to 9.0]
  Week 41 (Injection #6): number analyzed (Participants) | 1623 | 1608
  Week 41 (Injection #6) | 2.0 [-4.0 to 10.0] | 2.0 [-5.0 to 9.0]
  Week 49 (Injection #7): number analyzed (Participants) | 1465 | 1464
  Week 49 (Injection #7) | 3.0 [-4.0 to 10.0] | 2.0 [-5.0 to 10.0]
  Week 57 (Injection #8): number analyzed (Participants) | 1360 | 1358
  Week 57 (Injection #8) | 2.0 [-6.0 to 8.0] | 0.0 [-6.0 to 7.0]
  Week 65 (Injection #9): number analyzed (Participants) | 1207 | 1195
  Week 65 (Injection #9) | 2.0 [-4.0 to 10.0] | 2.0 [-5.0 to 10.0]
  Week 73 (Injection #10): number analyzed (Participants) | 1036 | 1036
  Week 73 (Injection #10) | 3.0 [-4.0 to 11.0] | 2.0 [-4.0 to 10.0]
  Week 81 (Injection #11): number analyzed (Participants) | 878 | 902
  Week 81 (Injection #11) | 3.0 [-4.0 to 11.0] | 2.0 [-5.0 to 10.0]
  Week 89 (Injection #12): number analyzed (Participants) | 746 | 759
  Week 89 (Injection #12) | 3.0 [-4.0 to 11.0] | 2.0 [-5.0 to 10.0]
  Week 97 (Injection #13): number analyzed (Participants) | 602 | 600
  Week 97 (Injection #13) | 3.0 [-5.0 to 12.0] | 2.0 [-4.0 to 11.0]
  Week 105 (Injection #14): number analyzed (Participants) | 461 | 482
  Week 105 (Injection #14) | 2.0 [-6.0 to 9.0] | 1.0 [-6.0 to 7.0]
  Week 113 (Injection #15): number analyzed (Participants) | 375 | 374
  Week 113 (Injection #15) | 4.0 [-4.0 to 11.0] | 2.0 [-4.0 to 10.0]
  Week 121 (Injection #16): number analyzed (Participants) | 298 | 290
  Week 121 (Injection #16) | 3.0 [-4.5 to 12.0] | 3.0 [-6.0 to 11.0]
  Week 129 (Injection #17): number analyzed (Participants) | 230 | 219
  Week 129 (Injection #17) | 2.0 [-5.5 to 11.0] | 2.0 [-6.0 to 10.0]
  Week 137 (Injection #18): number analyzed (Participants) | 168 | 148
  Week 137 (Injection #18) | 5.5 [-3.0 to 12.0] | 3.0 [-5.0 to 10.0]
  Week 145 (Injection #19): number analyzed (Participants) | 112 | 91
  Week 145 (Injection #19) | 4.0 [-4.0 to 13.0] | 2.0 [-6.0 to 11.0]
  Week 153 (Injection #20): number analyzed (Participants) | 59 | 55
  Week 153 (Injection #20) | 4.0 [-7.0 to 12.0] | 3.5 [-8.0 to 11.0]

11. Secondary Outcome: Changes in Fasting Glucose Levels From Baseline
Description: Changes in fasting glucose levels from baseline at week 57 and week 105 based on laboratory evaluations.
Time Frame: Assessed at weeks 57 and 105.
Population: Participants who were inappropriately enrolled are excluded. Inappropriately enrolled participants and participants with invalid ID due to duplicate screening or enrollment are excluded.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 2282 | 2284
mg/dL
  Week 57 | 1.0 [-5.0 to 7.0] | 0.0 [-6.0 to 6.0]
  Week 105 | 1.0 [-5.0 to 8.0] | 1.8 [-6.0 to 8.0]

12. Secondary Outcome: Changes in Fasting Lipid Profile From Baseline
Description: Changes in fasting lipid profile from baseline at week 57 and week 105 based on laboratory evaluations.
Time Frame: Assessed at weeks 57 and 105.
Population: Inappropriately enrolled participants and participants with invalid ID due to duplicate screening or enrollment are excluded.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cabotegravir | TDF/FTC
Number analyzed (Participants) | 2282 | 2284
mg/dL
  Total Cholesterol Week 57 | 1.0 [-15.0 to 16.0] | -10.0 [-26.0 to 6.2]
  Total Cholesterol Week 105 | 4.0 [-13.0 to 19.0] | -7.5 [-26.0 to 9.0]
  Trigylcerides Week 57 | 2.7 [-20.0 to 28.0] | 0.0 [-23.0 to 25.0]
  Trigylcerides Week 105 | 7.5 [-19.0 to 32.0] | 2.0 [-21.0 to 31.0]
  LDL Week 57 | 1.0 [-12.4 to 15.0] | -6.0 [-19.7 to 7.0]
  LDL Week 105 | 3.0 [-12.0 to 18.0] | -4.0 [-20.0 to 11.0]
  HDL Week57 | -0.2 [-6.0 to 5.0] | -3.0 [-9.0 to 3.0]
  HDL Week 105 | -0.9 [-6.8 to 5.0] | -3.0 [-9.0 to 2.6]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AE measured with onset date through participant's last study visit (up to 48 weeks after the last injection visit), or the date of DSMB decision to unblind all participants, whichever is earliest. Assessed at each visit (injections visits q 8 weeks and safety visits q 8 weeks)
Description: Includes the subset of subjects who received any study product, including those were subsequently deemed to be inappropriately enrolled.
Arm/Group | Cabotegravir | TDF/FTC
All-Cause Mortality (participants affected / at risk) | 4/2281 | 7/2285
Serious Adverse Events (participants affected / at risk) | 117/2281 | 109/2285
Other Adverse Events (participants affected / at risk) | 2103/2281 | 2114/2285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabotegravir (N=2281) | TDF/FTC (N=2285)
Any Event in SOC (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Any Event in SOC (Cardiac disorders) | 4 (4) | 6 (7)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Any Event in SOC (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Any Event in SOC (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Any Event in SOC (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Any Event in SOC (Gastrointestinal disorders) | 6 (6) | 7 (10)
Cannabinoid hyperemesis syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Any Event in SOC (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Any Event in SOC (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0)
Acute hepatitis B (Infections and infestations) | 2 (2) | 0 (0)
Acute hepatitis C (Infections and infestations) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Any Event in SOC (Infections and infestations) | 48 (50) | 38 (40)
Appendicitis (Infections and infestations) | 3 (3) | 9 (9)
Arthritis gonococcal (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Dengue fever (Infections and infestations) | 5 (5) | 3 (3)
Dengue haemorrhagic fever (Infections and infestations) | 2 (2) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 5 (5)
Hepatitis A (Infections and infestations) | 3 (4) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 2 (2)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphogranuloma venereum (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Secondary syphilis (Infections and infestations) | 0 (0) | 1 (1)
Shigella infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral pericarditis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Any Event in SOC (Injury, poisoning and procedural complications) | 13 (13) | 26 (26)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Any Event in SOC (Investigations) | 1 (1) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Any Event in SOC (Nervous system disorders) | 5 (5) | 4 (5)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 1 (1)
Any Event in SOC (Psychiatric disorders) | 23 (26) | 28 (32)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Borderline personality disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 6 (6)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Impulse-control disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 6 (6) | 6 (6)
Suicide attempt (Psychiatric disorders) | 8 (8) | 10 (11)
Any Event in SOC (Renal and urinary disorders) | 1 (1) | 2 (4)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (3)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Any Event in SOC (Vascular disorders) | 0 (0) | 3 (4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (3)
Vascular occlusion (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabotegravir (N=2281) | TDF/FTC (N=2285)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Any Event in SOC (Blood and lymphatic system disorders) | 33 (36) | 35 (40)
Cyclic neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4) | 7 (7)
Lymphocytic infiltration (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 15 (18) | 16 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3) | 0 (0)
Any Event in SOC (Cardiac disorders) | 8 (8) | 7 (7)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Any Event in SOC (Congenital, familial and genetic disorders) | 0 (0) | 3 (3)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Steatocystoma multiplex (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Thalassaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Any Event in SOC (Ear and labyrinth disorders) | 22 (24) | 24 (24)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 5 (5) | 5 (5)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear swelling (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 7 (8) | 6 (6)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Any Event in SOC (Endocrine disorders) | 2 (2) | 3 (3)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperprolactinaemia (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Any Event in SOC (Eye disorders) | 22 (30) | 20 (22)
Blepharitis (Eye disorders) | 1 (1) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Chorioretinopathy (Eye disorders) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 4 (4) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 2 (3) | 3 (3)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 2 (2) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Giant papillary conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 2 (2)
Hypermetropia (Eye disorders) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 2 (2) | 1 (1)
Ocular hyperaemia (Eye disorders) | 4 (5) | 2 (2)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Strabismus (Eye disorders) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 1 (1) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 26 (26) | 23 (24)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 24 (26) | 16 (17)
Anal fissure (Gastrointestinal disorders) | 20 (20) | 28 (31)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal inflammation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 6 (6) | 5 (6)
Anal skin tags (Gastrointestinal disorders) | 4 (4) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 3 (3) | 4 (4)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 4 (4) | 4 (5)
Any Event in SOC (Gastrointestinal disorders) | 450 (638) | 481 (706)
Aphthous ulcer (Gastrointestinal disorders) | 8 (8) | 10 (11)
Change of bowel habit (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 5 (5) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (14) | 16 (16)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 14 (14) | 11 (13)
Dental necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 111 (129) | 119 (152)
Dysbiosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 32 (38) | 31 (33)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 12 (12) | 12 (13)
Food poisoning (Gastrointestinal disorders) | 37 (38) | 41 (41)
Gastritis (Gastrointestinal disorders) | 29 (40) | 24 (27)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 (26) | 15 (15)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 7 (8)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 42 (45) | 44 (46)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (2) | 4 (5)
Lip exfoliation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 2 (2) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucous stools (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 22 (22) | 39 (48)
Odynophagia (Gastrointestinal disorders) | 15 (16) | 14 (14)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Parotid duct obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 2 (3)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 7 (7) | 15 (16)
Proctitis (Gastrointestinal disorders) | 14 (15) | 16 (17)
Rectal discharge (Gastrointestinal disorders) | 3 (3) | 3 (3)
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 5 (6)
Rectal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sialocele (Gastrointestinal disorders) | 0 (0) | 1 (3)
Steatorrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tooth deposit (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 11 (12) | 7 (7)
Toothache (Gastrointestinal disorders) | 28 (33) | 44 (48)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Uvulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (11) | 22 (22)
Adverse drug reaction (General disorders) | 0 (0) | 3 (3)
Adverse food reaction (General disorders) | 0 (0) | 1 (1)
Any Event in SOC (General disorders) | 229 (359) | 149 (174)
Application site pain (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 4 (4) | 4 (4)
Chest discomfort (General disorders) | 1 (2) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 4 (6) | 2 (2)
Cyst (General disorders) | 2 (2) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 2 (2)
Face oedema (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 5 (5) | 2 (2)
Fatigue (General disorders) | 31 (37) | 14 (14)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Fibrosis (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Hangover (General disorders) | 3 (3) | 2 (2)
Hernia (General disorders) | 0 (0) | 1 (1)
Induration (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 28 (38) | 20 (23)
Injury associated with device (General disorders) | 1 (1) | 2 (2)
Lithiasis (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 30 (44) | 16 (18)
Medical device site ulcer (General disorders) | 0 (0) | 1 (1)
Mucosal disorder (General disorders) | 0 (0) | 1 (1)
Nodule (General disorders) | 1 (1) | 3 (3)
Non-cardiac chest pain (General disorders) | 5 (5) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 4 (4)
Pain (General disorders) | 12 (13) | 7 (7)
Peripheral swelling (General disorders) | 1 (1) | 2 (2)
Polyp (General disorders) | 1 (1) | 1 (1)
Puncture site pain (General disorders) | 0 (0) | 1 (1)
Puncture site swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 121 (186) | 62 (69)
Swelling face (General disorders) | 1 (1) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 1 (1)
Xerosis (General disorders) | 1 (1) | 0 (0)
Any Event in SOC (Hepatobiliary disorders) | 16 (19) | 14 (24)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Deficiency of bile secretion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic fibrosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 3 (3)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 (8) | 5 (12)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to animal (Immune system disorders) | 1 (1) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 1 (1)
Allergy to chemicals (Immune system disorders) | 0 (0) | 1 (1)
Any Event in SOC (Immune system disorders) | 59 (64) | 53 (54)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 6 (6) | 3 (3)
Food allergy (Immune system disorders) | 14 (16) | 7 (7)
Hypersensitivity (Immune system disorders) | 13 (15) | 11 (12)
Jarisch-Herxheimer reaction (Immune system disorders) | 0 (0) | 2 (2)
Mite allergy (Immune system disorders) | 0 (0) | 1 (1)
Multiple allergies (Immune system disorders) | 5 (5) | 3 (3)
Mycotic allergy (Immune system disorders) | 0 (0) | 2 (2)
Perfume sensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 18 (18) | 19 (19)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 8 (8) | 12 (12)
Abscess neck (Infections and infestations) | 1 (1) | 1 (1)
Abscess of eyelid (Infections and infestations) | 0 (0) | 1 (1)
Abscess rupture (Infections and infestations) | 0 (0) | 1 (1)
Acanthamoeba keratitis (Infections and infestations) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 26 (27) | 43 (48)
Acute hepatitis B (Infections and infestations) | 3 (5) | 3 (3)
Acute hepatitis C (Infections and infestations) | 7 (7) | 6 (6)
Acute sinusitis (Infections and infestations) | 8 (8) | 9 (9)
Amoebic dysentery (Infections and infestations) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 5 (6) | 9 (10)
Anal candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Anal chlamydia infection (Infections and infestations) | 248 (297) | 267 (326)
Anal fistula infection (Infections and infestations) | 0 (0) | 1 (1)
Anal fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 1 (1) | 1 (1)
Anorectal human papilloma virus infection (Infections and infestations) | 9 (9) | 12 (12)
Any Event in SOC (Infections and infestations) | 1360 (3515) | 1344 (3456)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Arboviral infection (Infections and infestations) | 3 (3) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 5 (6) | 2 (2)
Bacterial infection (Infections and infestations) | 0 (0) | 3 (3)
Bacterial prostatitis (Infections and infestations) | 0 (0) | 1 (2)
Bacterial urethritis (Infections and infestations) | 9 (10) | 9 (9)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Balanitis candida (Infections and infestations) | 5 (5) | 3 (3)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Blastocystis infection (Infections and infestations) | 1 (1) | 2 (2)
Body tinea (Infections and infestations) | 7 (8) | 6 (6)
Bone abscess (Infections and infestations) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 2 (3) | 0 (0)
Bronchitis (Infections and infestations) | 28 (30) | 31 (32)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis viral (Infections and infestations) | 1 (1) | 3 (4)
Bullous impetigo (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 14 (14) | 11 (11)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (2)
Candida infection (Infections and infestations) | 1 (1) | 3 (3)
Candida urethritis (Infections and infestations) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 22 (24) | 11 (11)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 2 (2)
Chancroid (Infections and infestations) | 2 (2) | 2 (2)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Chikungunya virus infection (Infections and infestations) | 3 (3) | 4 (4)
Chlamydial infection (Infections and infestations) | 66 (77) | 66 (74)
Chronic hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 19 (19) | 24 (27)
Conjunctivitis bacterial (Infections and infestations) | 3 (3) | 2 (2)
Conjunctivitis viral (Infections and infestations) | 4 (4) | 3 (3)
Cryptosporidiosis infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 3 (3) | 2 (2)
Cystitis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 6 (6) | 6 (7)
Dengue haemorrhagic fever (Infections and infestations) | 1 (1) | 0 (0)
Dermatophytosis (Infections and infestations) | 8 (8) | 5 (5)
Diarrhoea infectious (Infections and infestations) | 12 (12) | 8 (8)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2)
Dysentery (Infections and infestations) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 13 (13) | 15 (19)
Ear infection bacterial (Infections and infestations) | 2 (2) | 1 (1)
Ear lobe infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 2 (2)
Enterovirus infection (Infections and infestations) | 4 (4) | 0 (0)
Epididymitis (Infections and infestations) | 6 (6) | 7 (7)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
External ear cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Eye infection (Infections and infestations) | 1 (1) | 1 (1)
Eye infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Eye infection gonococcal (Infections and infestations) | 1 (1) | 0 (0)
Eye infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 9 (9) | 5 (5)
Folliculitis (Infections and infestations) | 16 (17) | 14 (16)
Fungal infection (Infections and infestations) | 2 (2) | 3 (3)
Fungal skin infection (Infections and infestations) | 5 (5) | 7 (7)
Furuncle (Infections and infestations) | 15 (16) | 15 (16)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 83 (88) | 87 (94)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis cryptosporidial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 22 (22) | 14 (14)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 11 (11) | 4 (4)
Gastrointestinal protozoal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 2 (2) | 1 (1)
Genital candidiasis (Infections and infestations) | 6 (8) | 5 (5)
Genital herpes (Infections and infestations) | 23 (33) | 22 (36)
Genital herpes simplex (Infections and infestations) | 11 (12) | 10 (14)
Genital herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Genital infection (Infections and infestations) | 0 (0) | 1 (1)
Genital infection bacterial (Infections and infestations) | 0 (0) | 3 (3)
Genital infection fungal (Infections and infestations) | 3 (3) | 4 (4)
Genitourinary chlamydia infection (Infections and infestations) | 34 (37) | 23 (27)
Genitourinary tract gonococcal infection (Infections and infestations) | 21 (21) | 16 (17)
Giardiasis (Infections and infestations) | 4 (4) | 3 (3)
Gingival abscess (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 7 (7) | 9 (9)
Gonococcal infection (Infections and infestations) | 6 (6) | 2 (2)
Gonorrhoea (Infections and infestations) | 51 (60) | 49 (57)
Groin infection (Infections and infestations) | 1 (1) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 2 (2)
Helicobacter infection (Infections and infestations) | 2 (2) | 3 (3)
Helminthic infection (Infections and infestations) | 2 (2) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis syphilitic (Infections and infestations) | 0 (0) | 1 (1)
Herpes dermatitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 14 (19) | 10 (13)
Herpes virus infection (Infections and infestations) | 1 (1) | 3 (3)
Herpes zoster (Infections and infestations) | 7 (7) | 12 (12)
Hordeolum (Infections and infestations) | 17 (17) | 19 (19)
Impetigo (Infections and infestations) | 2 (2) | 4 (4)
Infected bite (Infections and infestations) | 2 (2) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infection parasitic (Infections and infestations) | 2 (2) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 5 (5)
Infectious thyroiditis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 62 (64) | 63 (65)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 3 (3) | 3 (3)
Laryngitis viral (Infections and infestations) | 0 (0) | 1 (1)
Latent syphilis (Infections and infestations) | 56 (58) | 50 (54)
Latent tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Lice infestation (Infections and infestations) | 3 (3) | 6 (6)
Localised infection (Infections and infestations) | 3 (3) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Lymphadenitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Lymphogranuloma venereum (Infections and infestations) | 4 (4) | 6 (6)
Malassezia infection (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 1 (1)
Measles (Infections and infestations) | 2 (2) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 2 (3) | 1 (1)
Mononucleosis syndrome (Infections and infestations) | 2 (2) | 1 (1)
Mumps (Infections and infestations) | 6 (6) | 2 (2)
Mycoplasma genitalium infection (Infections and infestations) | 1 (1) | 1 (1)
Myringitis (Infections and infestations) | 0 (0) | 1 (1)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 295 (421) | 273 (380)
Onychomycosis (Infections and infestations) | 13 (14) | 11 (11)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 26 (29) | 24 (27)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Oral pustule (Infections and infestations) | 0 (0) | 1 (1)
Oral viral infection (Infections and infestations) | 1 (2) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 2 (2)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal gonococcal infection (Infections and infestations) | 33 (35) | 27 (29)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 7 (7) | 6 (8)
Otitis externa bacterial (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa fungal (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 7 (8) | 3 (3)
Otitis media acute (Infections and infestations) | 7 (9) | 2 (2)
Otitis media bacterial (Infections and infestations) | 4 (4) | 0 (0)
Otitis media viral (Infections and infestations) | 1 (1) | 0 (0)
Papilloma viral infection (Infections and infestations) | 7 (7) | 4 (4)
Parasitic gastroenteritis (Infections and infestations) | 5 (5) | 9 (10)
Paronychia (Infections and infestations) | 9 (9) | 8 (8)
Parotitis (Infections and infestations) | 1 (2) | 3 (3)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Pericoronitis (Infections and infestations) | 0 (0) | 2 (2)
Periodontitis (Infections and infestations) | 2 (2) | 2 (2)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 2 (2)
Pharyngeal chlamydia infection (Infections and infestations) | 11 (11) | 5 (5)
Pharyngitis (Infections and infestations) | 104 (124) | 89 (101)
Pharyngitis bacterial (Infections and infestations) | 9 (9) | 8 (8)
Pharyngitis streptococcal (Infections and infestations) | 46 (52) | 29 (34)
Pharyngotonsillitis (Infections and infestations) | 6 (6) | 8 (9)
Pilonidal cyst (Infections and infestations) | 2 (4) | 4 (4)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 12 (12) | 11 (11)
Pneumonia bacterial (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 2 (2) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3) | 2 (2)
Primary syphilis (Infections and infestations) | 23 (25) | 23 (25)
Proctitis bacterial (Infections and infestations) | 1 (3) | 4 (4)
Proctitis chlamydial (Infections and infestations) | 34 (39) | 41 (47)
Proctitis gonococcal (Infections and infestations) | 200 (235) | 225 (256)
Proctitis herpes (Infections and infestations) | 3 (5) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Pulpitis dental (Infections and infestations) | 2 (2) | 4 (4)
Puncture site infection (Infections and infestations) | 1 (1) | 0 (0)
Purulent discharge (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 3 (3) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 4 (4)
Rhinitis (Infections and infestations) | 26 (35) | 18 (22)
Rocky mountain spotted fever (Infections and infestations) | 0 (0) | 1 (1)
Root canal infection (Infections and infestations) | 2 (2) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 2 (2)
Secondary syphilis (Infections and infestations) | 26 (26) | 31 (31)
Severe acute respiratory syndrome (Infections and infestations) | 1 (1) | 2 (2)
Sexually transmitted disease (Infections and infestations) | 4 (4) | 5 (5)
Shigella infection (Infections and infestations) | 0 (0) | 1 (2)
Sialoadenitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 44 (50) | 47 (52)
Sinusitis bacterial (Infections and infestations) | 4 (6) | 15 (15)
Skin bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 3 (3)
Staphylococcal infection (Infections and infestations) | 2 (2) | 3 (3)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 3 (3)
Streptococcal infection (Infections and infestations) | 0 (0) | 2 (2)
Strongyloidiasis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 12 (13) | 7 (9)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 3 (3)
Syphilis (Infections and infestations) | 187 (203) | 198 (219)
Syphilis anal (Infections and infestations) | 1 (1) | 0 (0)
Syphilis genital (Infections and infestations) | 2 (2) | 1 (1)
Tinea cruris (Infections and infestations) | 12 (16) | 11 (11)
Tinea infection (Infections and infestations) | 0 (0) | 3 (3)
Tinea pedis (Infections and infestations) | 4 (4) | 8 (8)
Tinea versicolour (Infections and infestations) | 8 (8) | 10 (10)
Tonsillitis (Infections and infestations) | 56 (63) | 59 (67)
Tonsillitis bacterial (Infections and infestations) | 23 (28) | 15 (16)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 15 (16) | 14 (18)
Tooth infection (Infections and infestations) | 15 (15) | 15 (15)
Tracheitis (Infections and infestations) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 2 (2)
Trichomoniasis (Infections and infestations) | 2 (2) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 176 (245) | 170 (223)
Upper respiratory tract infection bacterial (Infections and infestations) | 3 (3) | 2 (2)
Urethritis (Infections and infestations) | 51 (60) | 58 (63)
Urethritis chlamydial (Infections and infestations) | 56 (62) | 60 (66)
Urethritis gonococcal (Infections and infestations) | 64 (70) | 51 (61)
Urinary tract infection (Infections and infestations) | 25 (27) | 23 (24)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 3 (3)
Varicella (Infections and infestations) | 3 (3) | 3 (3)
Viral diarrhoea (Infections and infestations) | 6 (6) | 3 (3)
Viral infection (Infections and infestations) | 58 (62) | 48 (65)
Viral pharyngitis (Infections and infestations) | 14 (14) | 6 (6)
Viral rash (Infections and infestations) | 1 (1) | 0 (0)
Viral rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Viral sinusitis (Infections and infestations) | 3 (3) | 9 (11)
Viral tonsillitis (Infections and infestations) | 4 (4) | 7 (7)
Viral upper respiratory tract infection (Infections and infestations) | 59 (77) | 66 (77)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 9 (9) | 4 (4)
Wound infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 4 (4) | 5 (7)
Anal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 7 (7) | 6 (6)
Animal scratch (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Any Event in SOC (Injury, poisoning and procedural complications) | 286 (420) | 317 (437)
Arthropod bite (Injury, poisoning and procedural complications) | 7 (7) | 18 (20)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Back injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Burn oesophageal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Burns second degree (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Buttock injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 4 (6) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 16 (16) | 18 (20)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ear injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 17 (21) | 14 (16)
Exposure to contaminated air (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Eyelid injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Joint injury (Injury, poisoning and procedural complications) | 12 (14) | 8 (9)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 34 (39) | 36 (38)
Limb injury (Injury, poisoning and procedural complications) | 14 (15) | 20 (21)
Lip injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 33 (35) | 31 (36)
Nail avulsion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Penis injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Perineal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 5 (7)
Post procedural swelling (Injury, poisoning and procedural complications) | 9 (10) | 7 (8)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Prescribed overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 66 (73) | 71 (82)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Retinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 20 (22) | 10 (10)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 25 (28) | 24 (25)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 10 (11) | 8 (8)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 159 (189) | 192 (238)
Amylase increased (Investigations) | 148 (282) | 169 (292)
Any Event in SOC (Investigations) | 1892 (8346) | 1914 (9028)
Aspartate aminotransferase increased (Investigations) | 188 (216) | 197 (228)
Bilirubin conjugated increased (Investigations) | 1 (1) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 7 (8)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 89 (150) | 108 (169)
Blood calcium decreased (Investigations) | 3 (3) | 6 (6)
Blood calcium increased (Investigations) | 3 (3) | 4 (4)
Blood cholesterol increased (Investigations) | 41 (42) | 24 (24)
Blood creatine decreased (Investigations) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 4 (4) | 1 (1)
Blood creatine phosphokinase decreased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 484 (678) | 470 (682)
Blood creatinine decreased (Investigations) | 16 (17) | 15 (15)
Blood creatinine increased (Investigations) | 382 (711) | 428 (783)
Blood glucose decreased (Investigations) | 98 (119) | 103 (130)
Blood glucose increased (Investigations) | 199 (302) | 123 (190)
Blood phosphorus decreased (Investigations) | 90 (118) | 110 (152)
Blood phosphorus increased (Investigations) | 2 (2) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 6 (6)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure diastolic abnormal (Investigations) | 0 (0) | 1 (1)
Blood pressure diastolic increased (Investigations) | 3 (3) | 3 (3)
Blood pressure increased (Investigations) | 22 (29) | 19 (27)
Blood pressure systolic increased (Investigations) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 2 (2) | 0 (0)
Blood sodium increased (Investigations) | 2 (2) | 0 (0)
Blood testosterone decreased (Investigations) | 2 (2) | 1 (1)
Blood triglycerides increased (Investigations) | 31 (33) | 27 (30)
Blood uric acid increased (Investigations) | 2 (2) | 2 (2)
Creatinine renal clearance decreased (Investigations) | 1589 (4777) | 1671 (5351)
Creatinine renal clearance increased (Investigations) | 8 (8) | 6 (6)
Electrocardiogram QT prolonged (Investigations) | 3 (4) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 12 (16) | 19 (28)
Glucose urine present (Investigations) | 1 (1) | 2 (2)
HLA-B*27 positive (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3) | 3 (3)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 249 (457) | 260 (468)
Lipids increased (Investigations) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 60 (61) | 28 (28)
Lymphocyte count decreased (Investigations) | 12 (13) | 12 (13)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 22 (38) | 35 (61)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 6 (8) | 2 (2)
Protein urine (Investigations) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 2 (2)
Red blood cells urine (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 18 (26) | 41 (57)
White blood cell count decreased (Investigations) | 2 (9) | 2 (4)
Abnormal loss of weight (Metabolism and nutrition disorders) | 35 (44) | 63 (94)
Any Event in SOC (Metabolism and nutrition disorders) | 128 (169) | 160 (228)
Dairy intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Fructose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (2) | 4 (5)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 20 (28) | 18 (34)
Hyperlipasaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 23 (30) | 24 (28)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (10) | 17 (18)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lipid metabolism disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Overweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 8 (8) | 6 (6)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 247 (319) | 255 (325)
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 (44) | 44 (50)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 75 (90) | 88 (93)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Chondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 11 (11)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 58 (60) | 53 (63)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 11 (11)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (17) | 21 (23)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (8)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (8)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal retrolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (21) | 21 (24)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 (38) | 33 (39)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (2)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Penile wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 5 (5)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amputation stump pain (Nervous system disorders) | 0 (0) | 1 (1)
Any Event in SOC (Nervous system disorders) | 273 (388) | 270 (387)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (2)
Burning sensation (Nervous system disorders) | 0 (0) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 2 (3) | 2 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (5) | 2 (2)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cluster headache (Nervous system disorders) | 0 (0) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 11 (13) | 18 (20)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Essential tremor (Nervous system disorders) | 0 (0) | 1 (1)
Exertional headache (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 204 (275) | 195 (273)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 5 (5)
Lethargy (Nervous system disorders) | 0 (0) | 1 (3)
Loss of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 18 (27) | 13 (13)
Migraine with aura (Nervous system disorders) | 0 (0) | 2 (2)
Nerve compression (Nervous system disorders) | 1 (1) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 4 (4)
Presyncope (Nervous system disorders) | 3 (3) | 2 (2)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 6 (6) | 5 (5)
Seizure (Nervous system disorders) | 0 (0) | 4 (4)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 3 (3) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 8 (8) | 8 (10)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 24 (27) | 17 (19)
Abnormal dreams (Psychiatric disorders) | 3 (3) | 4 (4)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 2 (2) | 4 (4)
Adjustment disorder with depressed mood (Psychiatric disorders) | 4 (4) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 4 (4) | 2 (2)
Alcoholism (Psychiatric disorders) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 57 (62) | 45 (45)
Anxiety disorder (Psychiatric disorders) | 4 (4) | 3 (3)
Any Event in SOC (Psychiatric disorders) | 220 (285) | 196 (247)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 2 (2) | 6 (6)
Bipolar II disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 5 (5) | 4 (4)
Borderline personality disorder (Psychiatric disorders) | 1 (1) | 2 (2)
Bulimia nervosa (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 6 (6) | 9 (9)
Depression (Psychiatric disorders) | 66 (67) | 50 (52)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Discouragement (Psychiatric disorders) | 1 (1) | 1 (1)
Drug abuse (Psychiatric disorders) | 2 (2) | 0 (0)
Drug dependence (Psychiatric disorders) | 2 (2) | 4 (4)
Drug use disorder (Psychiatric disorders) | 2 (2) | 1 (1)
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Emotional distress (Psychiatric disorders) | 2 (2) | 0 (0)
Flashback (Psychiatric disorders) | 1 (1) | 0 (0)
Gambling disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Gender dysphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 2 (2) | 2 (2)
Grief reaction (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucinations, mixed (Psychiatric disorders) | 1 (1) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 49 (56) | 53 (56)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 2 (2) | 2 (2)
Libido decreased (Psychiatric disorders) | 6 (6) | 3 (3)
Major depression (Psychiatric disorders) | 8 (8) | 4 (4)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental fatigue (Psychiatric disorders) | 1 (1) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 2 (2) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 3 (3) | 4 (4)
Panic disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Panic reaction (Psychiatric disorders) | 1 (1) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 6 (6) | 4 (4)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Seasonal affective disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 2 (2) | 1 (1)
Substance abuse (Psychiatric disorders) | 2 (2) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 8 (8) | 11 (12)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Thinking abnormal (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Any Event in SOC (Renal and urinary disorders) | 77 (92) | 78 (85)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Choluria (Renal and urinary disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 26 (26) | 17 (17)
Glycosuria (Renal and urinary disorders) | 2 (2) | 6 (6)
Haematuria (Renal and urinary disorders) | 9 (9) | 16 (16)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 7 (9) | 10 (11)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 9 (10) | 11 (11)
Renal colic (Renal and urinary disorders) | 2 (2) | 1 (1)
Urethral discharge (Renal and urinary disorders) | 23 (27) | 15 (15)
Urethral syndrome (Renal and urinary disorders) | 2 (2) | 1 (1)
Urethritis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Any Event in SOC (Reproductive system and breast disorders) | 55 (67) | 54 (60)
Balanoposthitis (Reproductive system and breast disorders) | 7 (8) | 9 (10)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 5 (5) | 8 (8)
Erection increased (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Galactorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Genital burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital paraesthesia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Genital ulceration (Reproductive system and breast disorders) | 9 (9) | 8 (8)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nipple inflammation (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penile blister (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile discharge (Reproductive system and breast disorders) | 8 (8) | 7 (7)
Penile erosion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Penile rash (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Penile swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 6 (6) | 7 (7)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 2 (2) | 6 (6)
Scrotal dermatitis (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal ulcer (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Testicular cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Testicular oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 16 (18)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (5)
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 184 (249) | 194 (265)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (11)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (46) | 38 (42)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 12 (12)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal mucosal erosion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 41 (42) | 48 (50)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 32 (33) | 29 (35)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 24 (26)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 15 (16)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Small airways disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 18 (19) | 25 (27)
Acne cystic (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 5 (5)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 158 (185) | 189 (219)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 10 (10) | 10 (10)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 10 (11) | 11 (12)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 9 (10) | 12 (12)
Dermatitis papillaris capillitii (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lichen nitidus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 5 (5) | 9 (9)
Penile ulceration (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (14) | 10 (10)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 23 (28) | 23 (24)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Rash pruritic (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (5)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sea bather's eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 16 (18) | 19 (25)
Urticaria cholinergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Any Event in SOC (Social circumstances) | 1 (1) | 1 (1)
Impaired quality of life (Social circumstances) | 0 (0) | 1 (1)
Substance use (Social circumstances) | 1 (1) | 0 (0)
Any Event in SOC (Vascular disorders) | 39 (47) | 31 (37)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hyperaemia (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 35 (43) | 24 (29)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis superficial (Vascular disorders) | 0 (0) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
White coat hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT02720094/Prot_001.pdf
  • Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT02720094/SAP_002.pdf
  • Informed Consent Form (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT02720094/ICF_000.pdf